CLINICAL TRIAL: NCT00023348
Title: TBTC Study 23A: Pharmacokinetics of Intermittent Isoniazid and Rifabutin in USPHS Study 23: Treatment of HIV-Related Tuberculosis Using a Rifabutin-Based Regimen
Brief Title: TBTC Study 23A: Pharmacokinetics of Intermittent Isoniazid and Rifabutin in HIV-TB
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCHSTP-2173; 23A
Record Dates: First submitted 2001-09-06; First posted 2001-09-10 (Estimated); Last update posted 2005-09-13 (Estimated); Status verified 2005-09

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Tuberculosis; TB
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — Isoniazid; Rifabutin

INTERVENTIONS:
Drug: Isoniazid
Drug: Rifabutin

SUMMARY:
Primary Objectives:

1) To determine the proportion of patients with HIV-related tuberculosis who have abnormal pharmacokinetic parameters for isoniazid and rifabutin.

Secondary Objectives:

1. To determine risk factors for abnormal pharmacokinetic parameters for isoniazid and rifabutin.
2. To evaluate the correlation between pharmacokinetic parameters of isoniazid and rifabutin and the occurrence of toxicity attributed to antituberculous therapy.
3. To evaluate the correlation between pharmacokinetic parameters of isoniazid and rifabutin and the efficacy of TB therapy.
4. To define and correlate phenotypic INH acetylator status with the results of genotypic acetylator data obtained in the parent trial.

DETAILED DESCRIPTION:
This study will seek to enroll every eligible patient enrolled in TBTC Study 23. Consenting patients will be asked to undergo measurements of isoniazid (if receiving), rifabutin and 25-OH desacetyl rifabutin levels at a time point in the study when steady state rifabutin levels are expected to have been achieved (at least two weeks following the start of rifabutin).

ELIGIBILITY:
Inclusion:

1. Patient enrolled in TBTC Study 23
2. Informed consent

Exclusion:

1. Severe anemia (Hct <25%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 1999-07; Study Completion 2002-11

PRIMARY OUTCOMES:
To determine the proportion of patients with HIV-related tuberculosis who have abnormal pharmacokinetics of isoniazid and rifabutin.

SECONDARY OUTCOMES:
1) To determine risk factors for abnormal pharmacokinetics of isoniazid and rifabutin
2) To evaluate the correlation between pharmacokinetic parameters of isoniazid and rifabutin and the occurrence of toxicity attributed to antituberculous therapy.
3) To evaluate the correlation between pharmacokinetic parameters of isoniazid and rifabutin and the efficacy of TB therapy.
4) To define and correlate phenotypic INH acetylator status with the results of genotypic acetylator data obtained in the parent trial.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Weiner, MD, Principal Investigator — Audie L. Murphy VA Medical Center, San Antonio TX
Locations (23):
- United States (20):
  - Central Arkansas Veterans Health System, Little Rock, Arkansas
  - LA County/USC Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Denver Department of Public Health and Hospitals, Denver, Colorado
  - Washington, D.C. VAMC, Washington D.C., District of Columbia
  - Chicago VA Medical Center (Lakeside), Chicago, Illinois
  - Hines VA Medical Center, Hines, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - New Jersey Medical School, Newark, New Jersey
  - New York University School of Medicine, New York, New York
  - Columbia University/Presbyterian Medical Center, New York, New York
  - Harlem Hospital Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Nashville VA Medical Center, Nashville, Tennessee
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Thomas Street Clinic, Houston, Texas
  - Audi L. Murphy VA Hospital, San Antonio, Texas
  - Seattle King County Health Department, Seattle, Washington
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Montreal Chest Institute McGill University, Montreal, Quebec

REFERENCES:
- [Result] Weiner M, Benator D, Burman W, Peloquin CA, Khan A, Vernon A, Jones B, Silva-Trigo C, Zhao Z, Hodge T; Tuberculosis Trials Consortium. Association between acquired rifamycin resistance and the pharmacokinetics of rifabutin and isoniazid among patients with HIV and tuberculosis. Clin Infect Dis. 2005 May 15;40(10):1481-91. doi: 10.1086/429321. Epub 2005 Apr 14. PMID 15844071
- See also: (Click here for more information about the Tuberculosis Trials Consortium (TBTC) — http://www.cdc.gov/nchstp/tb/tbtc/